CLINICAL TRIAL: NCT07156240
Title: Impact of Two Short Behavioral Theory-Driven Professional Training Programs Targeting Attendance in Fitness Centers
Brief Title: Professional Training Programs Targeting Attendance in Fitness Centers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo Lusófona (Other)
Responsible Party: Principal Investigator, Diogo Teixeira, Professor, Grupo Lusófona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrupoLusofona
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-08

CONDITIONS: Exercise Frequency
Keywords: exercise; affect; motivation; adherence; frequency
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): FITT-VP 2025 training course
  Interventions: Other: Control group
- Experimental I (SDT) (Experimental): SDT-based training course
  Interventions: Behavioral: Experimental I (SDT)
- Experimental II (hedonic) (Experimental): Hedonic-based training course
  Interventions: Behavioral: Experimental II (Hedonic)

INTERVENTIONS:
Behavioral: Experimental I (SDT) — SDT-based course aiming to inmprove professionals operational interpersonal qualities
  Arms: Experimental I (SDT)
Behavioral: Experimental II (Hedonic) — Hedonic-based course aiming to inmprove professionals operational interpersonal qualities
  Arms: Experimental II (hedonic)
Other: Control group — FITT-VP bases course aiming to improve exercise prescription
  Arms: Control group

SUMMARY:
Over recent decades, leading theories of human behavior have been applied across various physical activity (PA) settings, yielding mixed results. While they have provided some valuable insights, they have largely failed to achieve one central aim - to help foster sustained, population-wide increases in PA (Albarracín et al., 2024; Ekkekakis & Zenko, 2016; Pratt et al., 2020; Rhodes et al., 2019). This gap has prompted concern, as these theories, despite some support for their assumptions, have not translated into meaningful and lasting behavior change. Some have criticized them for their overarching dependency on the decisional balance one may perform given the right set of conditions (e.g., supportive social environments; benefits vs. barriers dyad; self-efficacy appraisal) (Conn et al., 2011; Ekkekakis, 2017; Rhodes et al., 2019); others have pointed to an astonishing lack of experimental efforts testing the expression of those theoretical assumptions (Ekkekakis et al., 2019; Manninen et al., 2022; Ntoumanis & Moller, 2025), leaving researchers, policymakers and stakeholders (and the theories) hostage to cross-sectional and longitudinal evidence. Either way, new approaches and experimental efforts to address the challenge of supporting PA practices are warranted and urgent.

Three of the most studied motivational theories in PA contexts over the last decades are the Theory of Planned Behavior (Ajzen, 1991), Self-Determination Theory (Deci & Ryan, 1985), and the Transtheoretical Model (Prochaska & DiClemente, 1984) (Ntoumanis et al., 2018; Simpson et al., 2025). Without minimizing their usefulness and robust body of evidence, they fall into the category of theories that have struggled, to date, to demonstrate moderate or large effects in programs aiming to improve exercise-related behavior based on their assumptions. Naturally, the complexity of each theory or model brings several challenges that undermine the extent to which we can confidently attribute any limited effect observed in an experimental study solely to the theory's inability to express its assumptions. As such, despite decades of research grounded in several (conceptually) well-established behavioral theories, there remains a need to test their assumptions through experimental approaches and, complementarily - or if necessary, alternatively - to explore new avenues for inquiry and theoretical development (Simpson et al., 2025).

To this end, the present study will address this issue experimentally using two theoretical approaches. The first approach is grounded in a well-established theory of human motivation, Self-Determination Theory (SDT), which offers numerous recommendations for its potential application, particularly in promoting positive impacts on exercise adherence. The second approach is structured in alignment with the general principles of hedonic theory, a recently revitalized approach to the understanding of Human behavior, focusing on the promotion of pleasurable responses during exercise.

ELIGIBILITY:
Inclusion Criteria:

Professionals

- All exercise professionals in the three clubs

Exercisers

* > 18 years old
* All exercisers enrolled in the three clubs
* A subsample of the first 174 voluntaries participating in the study and enrolled in the three clubs after September 1st

Exclusion Criteria:

* Expulsion of the clubs due to internal rules violation or other decision independent of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Club attendance | Collected on the last day of each month, and averaged after a one-year period (September 1st to August 31st)
  Club attendance during a one-year period collected with the turstile digital system

SECONDARY OUTCOMES:
Attrition rate | Number of total cancellations or dropouts for each month, collected through the turstile digital record and club payment system, summed throughout 12 months
  Attrition rate calculated through the number of cancellations or dropouts / total number of new members × 100 in a one-year period
Exercise habit measured with the Self-reported behavioral automaticity index (SRBAI) - Baseline | Baseline; after club enrollment, in the first two weeks of September 2025, at any given time
  Automaticity for exercise practice measured with the Self-reported behavioral automaticity index (SRBAI)
Exercise habit measured with the Self-reported behavioral automaticity index (SRBAI) - 6 months | After 6 months of enrollment; first two weeks of February, at any given time
  Automaticity for exercise practice measured with the Self-reported behavioral automaticity index (SRBAI)
Exercise habit measured with the Self-reported behavioral automaticity index (SRBAI) - 12 months | After 12 months, during the last week of August 2026, at any given time
  Automaticity for exercise practice measured with the Self-reported behavioral automaticity index (SRBAI)
Initial behavioral intention to continue exercising; the intention to exercise questionnaire - Baseline | Baseline; after club enrollment, in the first two weeks of September 2025, at any given time
  Behavioral intention as defined by the theory of planned behavior with the intention to exercise questionnaire
Behavioral intention to continue exercising; the intention to exercise questionnaire - 6 months | After 6 months of enrollment; first two weeks of February, at any given time
  Behavioral intention as defined by the theory of planned behavior with the intention to exercise questionnaire
Behavioral intention to continue exercising; the intention to exercise questionnaire - 12 months | After 12 months, during the last week of August 2026, at any given time
  Behavioral intention as defined by the theory of planned behavior with the intention to exercise questionnaire
Exerciser basic psychological needs satisfaction and frustration; the BPNSFS questionnaire - Baseline | Baseline; after club enrollment, in the first two weeks of September 2025, at any given time
  Basic psychological needs satisfaction and frustration as defined by the Self-Determination Theory
Exerciser basic psychological needs satisfaction and frustration; the BPNSFS questionnaire - 6 months | After 6 months of enrollment; firts two weeks of February, at any given time
  Basic psychological needs satisfaction and frustration as defined by the Self-Determination Theory
Exerciser basic psychological needs satisfaction and frustration; the BPNSFS questionnaire - 12 months | After 12 months, during the last week of August 2026, at any given time
  Basic psychological needs satisfaction and frustration as defined by the Self-Determination Theory
Exerciser behavioral regulation; the BREQ-4 questionnaire - Baseline | Baseline; after club enrollment, in the first two weeks of September 2025, at any given time
  Exercise behavioral regulations as defined by the Self-Determination Theory
Exerciser behavioral regulation; the BREQ-4 questionnaire - 6 months | After 6 months of enrollment; firts two weeks of February, at any given time
  Exercise behavioral regulations as defined by the Self-Determination Theory
Exerciser behavioral regulation; the BREQ-4 questionnaire - 12 months | After 12 months, during the last week of August 2026, at any given time
  Exercise behavioral regulations as defined by the Self-Determination Theory
Exercise enjoyment measured with the Physical Activity Enjoyment Scale (PACES) - Baseline | Baseline; after club enrollment, in the first two weeks of September 2025, at any given time
  Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES)
Exercise enjoyment measured with the Physical Activity Enjoyment Scale (PACES) - 6 months | After 6 months of enrollment; firts two weeks of February, at any given time
  Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES)
Exercise enjoyment measured with the Physical Activity Enjoyment Scale (PACES) - 12 months | After 12 months, during the last week of August 2026, at any given time
  Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES)
Subjective exercise experience - Baseline | Baseline; after club enrollment, in the first two weeks of September 2025, at any given time
  The attraction-antipathy and the pleasure-displeasure assessed with the affective exercise experiences questionnaire (AFFEXX)
Subjective exercise experience - 6 months | After 6 months of enrollment; firts two weeks of February, at any given time
  The attraction-antipathy and the pleasure-displeasure assessed with the affective exercise experiences questionnaire (AFFEXX)
Subjective exercise experience - 12 months | After 12 months, during the last week of August 2026, at any given time
  The attraction-antipathy and the pleasure-displeasure assessed with the affective exercise experiences questionnaire (AFFEXX)

CONTACTS AND LOCATIONS:
Overall Officials: Diogo S. Teixeira, PhD, Principal Investigator — Lusófona University
Locations (1):
- People family club, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No